CLINICAL TRIAL: NCT00566826
Title: Perioperative Intervention to Improve Post-TKR Support and Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Patricia Franklin, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AR054479 (NIH); R01AR054479 (NIH); H 12601 (Other: University of Massachusetts Medical School)
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis; Arthroplasty, Replacement, Knee
Keywords: Physical Function; Total Knee Replacement; Physical Activity; Behavioral Support; Arthroplasty; Function; Self-Care
MeSH Terms: conditions — Osteoarthritis; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patient support treatment sessions
  Interventions: Behavioral: Patient support sessions
- 2 (Active Comparator): Treatment as usual
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Patient support sessions — Patient support sessions aim to enhance patient self-care for independent exercise and physical activity.
  Arms: 1
Behavioral: Treatment as usual — Treatment as usual includes standard care for TKR surgery rehabilitation.
  Arms: 2

SUMMARY:
Knee osteoarthritis is one of the most common causes of disability in older adults. Total knee replacement (TRK) surgery is often an effective solution when persistent pain does not sufficiently improve with non-surgical treatment. Although most TKR surgeries are a success, an estimated 15% to 30% of patients report no clinically significant improvement in function 12 months after a TKR. This study will evaluate the effectiveness of a patient support program in increasing physical function after a TKR surgery.

DETAILED DESCRIPTION:
Each year, more than 350,000 adults elect to have TKR surgery to eliminate knee pain and associated disabilities that persist despite ample medical treatment. Common knee problems of people who undergo TKR surgery include osteoarthritis, rheumatic diseases, and sudden or gradual joint injury. Most people who undergo TKR surgery experience immediate and significant decrease in pain, improved joint function, and increased physical activity. However, not all people who undergo TKR surgery report improvement, and there is no one factor that contributes to this variation in functional gain. With the rapid growth in the number of people electing to have TKR surgery and in the number of candidates eligible for TKR, optimal surgical results are both a clinical and public health priority. This study will evaluate the effectiveness of a patient support program emphasizing exercise and emotional health in increasing physical function after TKR surgery.

Participants in this study will be randomly assigned to a TKR patient support program or treatment as usual. The intervention patients will receive a program designed to complement the intensive physical rehabilitation period.

Sessions will aim to help participants enhance their self-management skills for behavior change.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for TKR surgery with one of University of Massachusetts Memorial Health Center's surgeons prior to study entry

Exclusion Criteria:

* TKR due to fracture, malignancy, infection, or failure of a previous knee replacement surgery
* Inability to return home during the rehabilitation period
* Co-existing conditions that would negate functional improvement with surgery and exercise
* TKR surgery scheduled on an emergency basis
* Scheduled for TKR surgeries of both knees at the same time
* Terminal illness with a life expectancy of less than 1 year
* Inability to provide informed consent due to dementia or cognitive impairment
* Planning another TKR or THR surgery within 6 months of study entry
* Unavailable to complete study procedures (i.e., will be out of the region during the rehabilitation period)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2008-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Physical function (SF36, WOMAC) | Measured at Months 6 and 12

SECONDARY OUTCOMES:
Physical activity and exercise | Measured at Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Patricia D. Franklin, MD, Principal Investigator — University of Massachusetts, Worcester; Milagros C. Rosal, PhD, Study Director — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Memorial Health Center; Arthritis and Total Joint Center, Worcester, Massachusetts, United States

REFERENCES:
- [Result] Ayers DC, Li W, Oatis C, Rosal MC, Franklin PD. Patient-reported outcomes after total knee replacement vary on the basis of preoperative coexisting disease in the lumbar spine and other nonoperatively treated joints: the need for a musculoskeletal comorbidity index. J Bone Joint Surg Am. 2013 Oct 16;95(20):1833-7. doi: 10.2106/JBJS.L.01007. PMID 24132356
- [Result] Zheng H, Rosal MC, Li W, Borg A, Yang W, Ayers DC, Franklin PD. A Web-Based Treatment Decision Support Tool for Patients With Advanced Knee Arthritis: Evaluation of User Interface and Content Design. JMIR Hum Factors. 2018 Apr 30;5(2):e17. doi: 10.2196/humanfactors.8568. PMID 29712620
- [Derived] Oatis CA, Johnson JK, DeWan T, Donahue K, Li W, Franklin PD. Characteristics of Usual Physical Therapy Post-Total Knee Replacement and Their Associations With Functional Outcomes. Arthritis Care Res (Hoboken). 2019 Sep;71(9):1171-1177. doi: 10.1002/acr.23761. PMID 30281207
- [Derived] Rosal MC, Ayers D, Li W, Oatis C, Borg A, Zheng H, Franklin P. A randomized clinical trial of a peri-operative behavioral intervention to improve physical activity adherence and functional outcomes following total knee replacement. BMC Musculoskelet Disord. 2011 Oct 7;12:226. doi: 10.1186/1471-2474-12-226. PMID 21981909